CLINICAL TRIAL: NCT05472844
Title: The Cohort Study of Pediatric Cataract
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2022KYPJ099
Record Dates: First submitted 2022-06-06; First posted 2022-07-25 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Cataract
Keywords: congenital cataract; traumatic cataract; complicated cataract; ocular structure parameters; surgical/vision recovery timing and strategies; postoperative adverse effects; psychologic and cognitive function; artificial intelligence
MeSH Terms: conditions — Capsule Opacification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The whole blood samples of participants and parents are collected and retained in our biobank for gene sequencing, hoping to explore the genetic factors in association with pathogenesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective-prospective bidirectional cohort study aims to observe ocular parameter changes, different surgical/vision recovery strategies and postoperative adverse effects among young children with cataract. The influence on psychology and cognitive function will be taken into consideration as well.

DETAILED DESCRIPTION:
Pediatric cataract, one of the leading causes of childhood blindness globally, is complex and of great difficulty in treatment. Pediatric patients with cataract (congenital, traumatic or complicated) are enrolled. In this study, investigators will compare ocular parameter changes, different surgical/vision timing or recovery strategies and adverse effects among young children （age < 18 yo）before and after cataract surgery. The influence on psychology and cognitive function will be taken into consideration as well. The whole blood samples of participants and parents are collected and retained in our biobank for gene sequencing, hoping to explore the genetic factors in association with pathogenesis. For children received cataract surgery, samples of partial anterior capsular tissue and 1 ml aqueous humor were collected during operation for further analysis. Multimodal artificial intelligence analyses are performed to establish accurate diagnosis/treatment scheme and disease prediction model.

ELIGIBILITY:
Inclusion Criteria:

* aged < 18 yo at the 1st visit unilateral or bilateral cataract agree to participant in this study and sign the informed consent

Exclusion Criteria:

* adults

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a retrospective-prospective bidirectional cohort study. Patients aged < 18 yo at the 1st visit are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity changes | Baseline and through study completion, an average of 1 year
  Best-corrected visual acuity changes are measured by visual acuity charts (Teller/Lea symbol/ETDRS chart) every 1 year at scheduled time
Intraocular pressure changes | Baseline and through study completion, an average of 1 year
  Intraocular pressures are measured by NCT machine
Refractive power changes | Baseline and through study completion, an average of 1 year
  Refractive power are measured at baseline and every visit at least every 1 year
Ocular biological measurements changes | Baseline and through study completion, an average of 1 year
  Ocular biological measurements including axial length, corneal keratometry, anterior chamber angle/depth, corneal endothelial cell number and appearance
Incidence changes of postoperative complications | Baseline and through study completion, an average of 1 year
  Incidence of postoperative complications, such as glaucoma-related adverse, myopic shift, strabismus and anisometropia and so on

SECONDARY OUTCOMES:
Other factors changes | Baseline and through study completion, an average of 1 year
  Sleep, depression, cognitive function are measured by questionnaires. Self-Rating Scale of Sleep: minimum value-1 point, maximum value-50, and higher scores mean worse outcome. Hamilton Depression Scale: <7 points-normal, and higher scores mean worse outcome. Loewenstein Cognitive Assessment: for every question, minimum 1 point, and maximum 4 points. Higher scores mean worse outcomes.
BMI changes | Baseline and through study completion, an average of 1 year
  BMI is measured by technicians in every visit
Blood pressure changes | Baseline and through study completion, an average of 1 year
  Diastolic and systolic blood pressure are measured by technicians in every visit
Stereopsis changes | Baseline and through study completion, an average of 1 year
  Stereopsis is measured by Randot Stereotest
Optical coherence tomography (OCT) changes | Baseline and through study completion, an average of 1 year
  Retinal thickness is measured and analyzed by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solebo AL, Teoh L, Rahi J. Epidemiology of blindness in children. Arch Dis Child. 2017 Sep;102(9):853-857. doi: 10.1136/archdischild-2016-310532. Epub 2017 May 2. PMID 28465303
- [Background] Chak M, Wade A, Rahi JS; British Congenital Cataract Interest Group. Long-term visual acuity and its predictors after surgery for congenital cataract: findings of the British congenital cataract study. Invest Ophthalmol Vis Sci. 2006 Oct;47(10):4262-9. doi: 10.1167/iovs.05-1160. PMID 17003414
- [Background] Long E, Zhang X, Liu Z, Wu X, Tan X, Lin D, Cao Q, Chen J, Lin Z, Wang D, Li X, Li J, Wang J, Li W, Lin H, Chen W, Liu Y. Dynamic response to initial stage blindness in visual system development. Clin Sci (Lond). 2017 Jun 28;131(13):1515-1527. doi: 10.1042/CS20170234. Print 2017 Jul 1. PMID 28539328